CLINICAL TRIAL: NCT07174648
Title: Field Evaluation of a Novel Antigen Rapid Diagnostic Test for Plague in the Province of Ituri, DR Congo
Brief Title: Testing of a New Rapid Antigen Test for Plague in Ituri, Democratic Republic of the Congo.
Acronym: RAPIDIT
Status: Not yet recruiting | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: ANRS | Maladies infectieuses émergentes (Unknown); Institut Pasteur (Industry); Université Paris-Saclay (Other); Centre de Recherche en Maladies Tropicales de L'Ituri (CRMT) (Unknown); Institut National pour la Recherche Biomedicale (INRB) (Unknown)
Responsible Party: Sponsor
Other Study IDs: RAPIDIT
Record Dates: First submitted 2025-09-08; First posted 2025-09-16 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Plague; Bubonic; Plague, Skin; Plague, Pneumonic
Keywords: Plague; Bubonic Plague; Pneumonic Plague; Ituri; DRC; Antigen rapid diagnostic test
MeSH Terms: conditions — Plague

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bubonic Aspirate, Sputum, Saliva, Gingival sulcus swabs, venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1: Cross-sectional Nested test-negative case-control study

SUMMARY:
This study is being done to learn more about the disease in Ituri and to evaluate a new rapid test that may help doctors find the disease more quickly. This research includes characterisation of clinical presentations and pathology of plague, as well as identification of circumstances that may increase the risk of infection. Biological samples collected include blood, mouth swab, saliva, a bubo aspirate and a sputum sample (the latter only in case of plague in the lungs). These samples will be used to test the performance of the new rapid study test.

DETAILED DESCRIPTION:
Plague is a life-threatening infection caused by the bacterium Yersinia pestis, which is highly endemic in the Ituri Province of the Democratic Republic of Congo (DRC) and associated with recurrent risks of regional epidemic spread. Clinical presentations (bubonic and/or pulmonary) and outcome remain poorly characterised in this area, and diagnostic accuracy is limited due to absence of a local bacteriology laboratory.

A novel lateral-flow immunochromatographic duplex rapid diagnostic test (RDT) has been developed for plague, which detects both F1 and LcrV proteins, and appears superior to the current RDT detecting only F1 antigens. This index RDT (called Duplex F1V) has shown promise in detecting Yersinia pestis in various sample types, including blood, bubo aspirates, and saliva in human patients.

Cross-sectional diagnostic accuracy study in clinical suspects of plague, comparing the results of Duplex F1V RDT (index assay), with PCR (polymerase chain reaction) positivity (as reference assay) on different biological fluids and assessment of clinical outcome at the end of treatment (at day 10-14).

Nested test-negative case-control study to identify risk factors and clinical predictors in PCR-confirmed plague cases, compared to PCR-negative suspects.

The study will take place in the Ituri province of DRC, the world's largest plague focus. Participants will be recruited in health centers and reference hospitals in the health areas of Rethy, Logo and Aru where the teams of the "Centre de Recherche en Maladies Tropicales" (CRMT) of Ituri are active. Individuals ≥5 years of age presenting at the sites with clinical suspicion of plague -as per national clinical case definitions- will be enrolled after informed consent and followed-up until treatment completion.

ELIGIBILITY:
Inclusion Criteria:

* All participants (aged ≥5 year old) within Rethy, Logo and Aru health zones, presenting with possible symptoms of bubonic and/or pneumonic plague according to WHO definition
* Willing to provide voluntary consent (or voluntary assent and parental consent in case of minors.

Exclusion Criteria:

* Participants not eligible, able, or willing to undergo study procedures
* Children <5 years of age
* Participants on antibiotic treatment ≥48h prior to recruitment

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People (> 5 years of age), living within Rethy, Logo and Aru health zones
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2029-01-02 (Estimated); Study Completion 2029-01-02 (Estimated)

PRIMARY OUTCOMES:
Duplex F1V RDT performance | 3 years
  Sensitivity, specificity, positive and negative predictive value of the Duplex F1V RDT results on different biological fluids, i.e. (1) gingival sulcus fluid, (2) saliva, (3) venous blood, (4) bubo aspirates and/or (5) sputum (depending on clinical presentation), as compared to positive PCR

IPD SHARING:
Plan to Share IPD: Undecided
Only anonymized individual participant data may be shared. Details are still under discussion with the relevant partners